CLINICAL TRIAL: NCT05302297
Title: A reTrOspective Study on Patient's Data From the French Cemiplimab Cohort ATU Programs Compared to Standard of Care in France
Brief Title: Comparative Efficacy of Cemiplimab to Historical Standard of Care in France
Acronym: TOSCA
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17334; U1111-1275-9937 (Registry Identifier: ICTRP)
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Cancer/Squamous Cell Carcinoma of Skin
MeSH Terms: conditions — Neoplasms | interventions — cemiplimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment Group (Cemiplimab): Patients treated with cemiplimab in monotherapy through the Cohort Temporary Authorization for Use (cATU) or patients included in the Nominative Temporary Authorization for Use( nATU) that evolved into the cATU and meeting the inclusion/exclusion criteria of the study.
  Interventions: Drug: Cemiplimab
- Control Group: Patients treated with other systemic treatments meeting the inclusion/exclusion criteria of the study who initiated at least one systemic treatment for advanced CSCC before start date of the cemiplimab nATU
  Interventions: Drug: Cemiplimab

INTERVENTIONS:
Drug: Cemiplimab — Pharmaceutical Form: Concentrate solution for injection for intravenous (IV) infusion Route of Administration: Intravenous (IV) infusion
  Other Names: SAR439684- Libtayo

SUMMARY:
Primary Objective:

-Assess the effectiveness of cemiplimab versus other available systemic therapies in patients up to 2018 or say historical system organ class (SOC) with metastatic or locally advanced cutaneous Squamous Cell Carcinoma (CSCC) who are not candidates for curative surgery or curative radiation, on overall survival (OS).

Secondary Objectives:

* Assess Progression Free Survival (PFS)
* To assess Duration of Response (DOR)
* To assess Objective Response Rate (ORR)
* To describe adverse events leading to treatment interruptions and deaths

DETAILED DESCRIPTION:
Study duration is approximately 9 months. For the Standard of Care Arm, data of the subjects evaluated between 01 Aug 2013 and 01 Aug 2018 was observed. For the Cemiplimab arm, data of the subjects evaluated between Aug 2018 and October 2019 was observed.

ELIGIBILITY:
Inclusion Criteria:

All patients:

* Adult 18 years of age or older
* With an unresectable locally advanced CSCC (who are not candidates for curative surgery or curative radiation therapy) or metastatic CSCC (nodal or distant)
* Subject alive at start data collection who has received information note and has not opposed to data collection OR

  * Subject who died before study initiation and who has not opposed to data collection for research purpose when he/she was alive

Treatment Group:

* Patient treated by cemiplimab in monotherapy through the cATU or patient included in the nATU that evolved into the cATU.
* With an Eastern Cooperative Oncology Group (ECOG) score of 0 or 1 at the time of cemiplimab initiation

Control Group:

* Patient treated by any systemic treatment initiated until August 1st , 2018 included
* With an ECOG score of 0 or 1 at the time of treatment initiation for at least one line of systemic therapy initiated from August 1st 2013 to August 1st 2018. The related treatment line must be among the 3 first systemic treatment lines for patients having initiated more than 3 lines.

Exclusion Criteria:

All patients:

- Patient treated by another anti- Programmed Cell Death Receptor-1 (PD1)

Control group:

-Patient subsequently treated with cemiplimab

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population for this study will be adult patients with metastatic or locally advanced CSCC who are not candidates for curative surgery or curative radiation and who received cemiplimab in monotherapy through the cATU or patient included in the nATU that evolved into the cATU (treatment group) and patients who initiated a systemic therapy as 1st, 2nd or 3rd line of treatment before the start of the cemiplimab nATU, i.e. initiated from August 1st 2013 to August 1st 2018 (control group) recruited from particpating sites in France. The study will aim to enroll approximately 250 patients in the cemiplimab group and 625 patients in the control group from up to 34 sites which included at least 4 patients in the cohort temporary authorization of use.
Sampling Method: Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | From patient advanced CSCC diagnosis date up to last medical record available on site or the end of the observation period (July 2022),whichever occurred first
  The difference OS between treatment and control groups expressed as a Hazard Ratio (HR). OS is the time between treatment initiation and the date of death from any cause. For participants who are alive at data cutoff collection, their survival time will be censored at the last date that they were known to be alive.

SECONDARY OUTCOMES:
Progression-Free Surivival (PFS) | From patient advanced CSCC diagnosis date up to last medical record available on site or the end of the observation period (July 2022),whichever occurred first
  Difference in PFS between interventional and control groups expressed as a HR. Defined as the time elapsed from date of first treatment intake to the date of documented recurrent or progressive disease reported by the Investigator or death due to any cause, whichever occurs first. Disease progression will be assessed by tumour response evaluation according to Investigator assessment. Tumour response will be evaluated per routine clinical practice as progressive/not progressive by the physian.
Duration of Response (DOR) | From patient advanced CSCC diagnosis date up to last medical record available on site or the end of the observation period (July 2022),whichever occurred first
  Defined as the time elapsed between the first reported objective response (complete or partial response) and the first date of recurrent or progressive disease or death due to any cause, whichever occurs first. Tumour response will be evaluated per routine clinical practice by the physician.
Objective Response Rate (ORR) | From patient advanced CSCC diagnosis date up to last medical record available on site or the end of the observation period (July 2022),whichever occurred first
  Defined as the proportion of participants who achieve partial or complete response from the start of the study treatment. The ORR will be assessed by tumour response evaluation according to Investigator assessment. Tumour response will be evaluated per routine clinical practice by the physician)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- France, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org